CLINICAL TRIAL: NCT03809364
Title: Supporting Treatment for Anti-Retroviral Therapy (START) Together: Development of a Couple-based Medication Adherence Intervention for HIV-positive Women and Their Male Partners in Sweetwaters, South Africa
Brief Title: Pilot Test of a Couple-Based Medication Adherence Intervention for HIV-Positive Women and Their Male Partners in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: Human Sciences Research Council (Other Government); University of Washington (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 395623
Record Dates: First submitted 2019-01-09; First posted 2019-01-18 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Human Immunodeficiency Virus
Keywords: Couple-based intervention; Antiretroviral therapy; South Africa
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- START Together (Experimental): Couples randomized to START Together will receive the manualized treatment to enhance women's medication adherence. The treatment is 5 sessions in length and conducted weekly. Sessions are 60 - 75 minutes. Couples have the option of completing up to 3 additional booster sessions. Total treatment therefore ranges between 5 to 8 sessions.
  Interventions: Behavioral: START Together
- Standard of Care (SOC) (No Intervention): Couples randomized to SOC will receive referrals to local HIV clinics to support medication adherence (for women) or other HIV-related issues (for men).

INTERVENTIONS:
Behavioral: START Together — Behavioral intervention using a cognitive behavioral couple therapy (CBCT) framework designed to improve the couple's communication and problem-solving behavior.
  Arms: START Together

SUMMARY:
The purpose of this study is to collect quantitative data related to developing and testing a couple-based intervention (CBI) for HIV-positive women's medication adherence in the region of Kwazulu-Natal, South Africa. The CBI, called START (Supporting Treatment for Anti-Retroviral Therapy) Together, will be a manualized intervention focused on women's ART adherence and enhancing the couple's communication and problem-solving behavior. The study focuses on implementation outcomes (feasibility, acceptability, and fidelity) and preliminary efficacy outcomes (women's ART adherence, men's engagement in HIV care, and the couple's relationship functioning), which will be compared to a control condition of referrals to usual HIV care.

DETAILED DESCRIPTION:
South Africa (SA) has one of the highest global HIV burdens with clear gender disparities. For men, 57% of HIV-related deaths occur among persons who have never sought HIV care. Women, in comparison, have high rates of HIV testing and are linked to care through antenatal services, but only 45% are virally suppressed on antiretroviral therapy (ART). Thus, tailored interventions for HIV are needed. In order to end the AIDS epidemic, the ambitious "90-90-90" goal was developed by UNAIDS to test, treat, and maintain medication adherence for 73% of HIV-positive individuals. Separate gender-specific interventions have been developed along the HIV care cascade to treat the different needs of men and women. However, no study to date has used one intervention to concurrently meet the unique HIV-related needs for women and men. Couple-based interventions (CBIs) can achieve this goal. CBIs are more efficacious than interventions delivered to individuals in enhancing a number of HIV protective behaviors. HIV is also primarily transmitted in the context of stable heterosexual relationships in sub-Saharan Africa; about 50% of new infections occur in serodiscordant relationships, making the use of a CBI especially relevant. The purpose of this study is to strengthen the HIV care cascade in SA by developing a CBI that concurrently addresses the needs of women and men to meet the UNAIDS' HIV goals. This study will be conducted in the province of KwaZulu-Natal, SA. HIV-positive women who are in a heterosexual relationship and non-adherent to ART will be recruited to participate in the study with their male partners. Twenty couples will be recruited and randomized to either receive the START Together program or to the control condition and followed for 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Both partners aged 18 or over
* HIV-positive woman diagnosed ≥ 3 months prior to study entry
* HIV-positive woman demonstrates difficulty with HIV treatment engagement, defined as either self-reported ART adherence difficulties, evidence of missed clinic visits over the past year (collected from medical records), or evidence of being not virally suppressed (≥ 50 copies/mL) in the past year
* In a committed, heterosexual, monogamous romantic relationship for at least 6 months
* Both partners willing to participate in treatment to support women's ART adherence
* Both partners reside in Vulindlela, or neighboring community, KwaZulu-Natal, South Africa
* Willing to have intervention sessions audio-recorded (if randomized to the intervention group)
* Able to comfortably communicate in either isiZulu or English

Exclusion Criteria:

* Report of moderate or severe relationship violence past year
* Either partner previously participated in a couple-based HIV prevention or treatment program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — HIV-positive women are the target study participants. They will participate in treatment with their male partners.
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Percentage of couples assigned to START Together who agree to enroll in the intervention | Approximately 8 weeks post-randomization
  Feasibility of START Together intervention
Average score on the 14-item Applied Mental Health Research group's feasibility subscale | Approximately 8 weeks post-randomization
  Feasibility of START Together intervention. Higher scores indicate greater feasibility.
Percentage of couples assigned to START Together who complete all treatment sessions | Approximately 8 weeks post-randomization
  Acceptability of START Together intervention
Average number of START Together sessions attended | Approximately 8 weeks post-randomization
  Acceptability of START Together intervention
Average score on the 15-item Applied Mental Health Research group's acceptability subscale | Approximately 8 weeks post-randomization
  Acceptability of START Together intervention. Higher scores indicate greater acceptability.
Average percentage of session content and process items that were completed correctly by the interventionist | Approximately 8 weeks post-randomization
  START Together intervention fidelity

SECONDARY OUTCOMES:
Viral suppression for women | Change from baseline assessment to approximately 12 weeks post-randomization
  Viral load in dried blood spots or based on clinic records (past 30 days)
HIV medication adherence for women | Change from baseline assessment to approximately 8 weeks post-randomization
  Self-report using the Ira Wilson adherence measure. Higher scores indicate better adherence
HIV medication adherence for women | Change from baseline assessment to approximately 12 weeks post-randomization
  Self-report using the Ira Wilson adherence measure. Higher scores indicate better adherence
Engagement in HIV care for men | Change from baseline assessment to approximately 12 weeks post-randomization
  Dichotomous engagement in care (yes/no) will be measured by clinic records review. If clinic records are unavailable, participant self-report will be used.
Relationship functioning (women and men) | Change from baseline assessment to approximately 8 weeks post-randomization
  Total score and subscales (relationship building, open communication, and couple-level problem-solving) of the South Africa Healthy Relationships Questionnaire. Higher scores indicate better relationship functioning.
Relationship functioning (women and men) | Change from baseline assessment to approximately 12 weeks post-randomization
  Total score and subscales (relationship building, open communication, and couple-level problem-solving) of the South Africa Healthy Relationships Questionnaire. Higher scores indicate better relationship functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Sciences Research Council, Pietermaritzburg, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crepaz N, Tungol-Ashmon MV, Vosburgh HW, Baack BN, Mullins MM. Are couple-based interventions more effective than interventions delivered to individuals in promoting HIV protective behaviors? A meta-analysis. AIDS Care. 2015;27(11):1361-6. doi: 10.1080/09540121.2015.1112353. Epub 2015 Nov 25. PMID 26608175
- [Background] Anglemyer A, Horvath T, Rutherford G. Antiretroviral therapy for prevention of HIV transmission in HIV-discordant couples. JAMA. 2013 Oct 16;310(15):1619-20. doi: 10.1001/jama.2013.278328. PMID 24129466
- [Background] Bor J, Rosen S, Chimbindi N, Haber N, Herbst K, Mutevedzi T, Tanser F, Pillay D, Barnighausen T. Mass HIV Treatment and Sex Disparities in Life Expectancy: Demographic Surveillance in Rural South Africa. PLoS Med. 2015 Nov 24;12(11):e1001905; discussion e1001905. doi: 10.1371/journal.pmed.1001905. eCollection 2015 Nov. PMID 26599699